CLINICAL TRIAL: NCT04763070
Title: Effect of Ciprofloxacin on Seizure Frequency in Patients With Drug-resistant Epilepsy
Brief Title: Ciprofloxacin in Drug-resistant Epilepsy
Acronym: CIDRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mazandaran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Nasim Tabrizi, Associate professor of neurology, Mazandaran University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5210
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Epilepsy Intractable
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ciprofloxacin (Other)
  Interventions: Drug: Ciprofloxacin Oral Product

INTERVENTIONS:
Drug: Ciprofloxacin Oral Product — The first stool sample will be taken before treatment and the second one will be taken in day 5 to 7 after treatment initiation. Treatment includes ciprofloxacin tablet 500mg twice a day for 5 days.

SUMMARY:
This study aims to investigate the effect of a short-term prescription of ciprofloxacin on intestinal microbial pattern and seizure frequency of patients with drug-resistant epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Drug-resistant epilepsy with frequency of at least 2 seizure/Week
* Acceptance of patients or his/her guardian (Signing informed consent)

Exclusion Criteria:

* Hypersensitivity to ciprofloxacin or other fluoroquinolones
* History of tendon, renal, hepatic or cerebrovascular disease, organ transplantation or myasthenia gravis
* Usage of medications with interaction to ciprofloxacin
* No reliable contraception
* Pregnancy or breastfeeding
* Being under treatment with corticosteroid
* Usage of antibiotics in recent 2 months or need to use it during the study
* Patients who are candidate for epilepsy surgery or other nonmedical treatments
* Change in anti-seizure medications (ASMs) during recent month
* Patients who will need changes in ASMs dose during study

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Changes in seizure frequency registered in questionnaire | 4 weeks
  Comparison of seizure frequency in 4th week with the frequency at the start of the study.
Changes in quantity of microbial DNA extracted from stool samples by AccuPrep Stool DNA extraction Kit | 7 days
  Comparison of quantity of extracted microbial DNA in stool sample taken at day5-7 with the sample taken at the start of the study
Changes in microbial burden of stool samples using Absolute real time polymerase chain reaction (PCR) | 7 days
  Comparison of microbial burden of stool samples taken at day5-7 with the sample taken at the start of the study

SECONDARY OUTCOMES:
Changes in seizure frequency registered in questionnaire | 12 weeks
  Comparison of seizure frequency in 12th week with the frequency at the start of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Bu Ali Sina hospital, Sari, Mazandaran, Iran

IPD SHARING:
Plan to Share IPD: No